CLINICAL TRIAL: NCT04348162
Title: Food Anthocyanins and Flavanols as a Strategy for a Healthy Ageing: Cardiovascular Health and Cognitive Performance
Acronym: POLYAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Principal Investigator, Spanish National Research Council, PhD, National Research Council, Spain
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AGL2016-76832-R
Record Dates: First submitted 2020-03-26; First posted 2020-04-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2020-04

CONDITIONS: Healthy Aging

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cocoa Flavanols (Active Comparator): Cocoa is taken every day for 10-12 weeks.
  Interventions: Other: Cocoa flavanols and berries anthocyanins
- Berries anthocyanins (Active Comparator): Red-berries are taken every day for 10-12 weeks.
  Interventions: Other: Cocoa flavanols and berries anthocyanins
- Cocoa flavanols plus berries anthocyanins (Active Comparator): Cooa and red-berries are taken every day for 10-12 weeks.
  Interventions: Other: Cocoa flavanols and berries anthocyanins
- Control (No Intervention): Normal diet for 10-12 weeks

INTERVENTIONS:
Other: Cocoa flavanols and berries anthocyanins — Effect of cocoa flavanols and berries anthocyanins on cardiovascular and cognitive health
  Arms: Berries anthocyanins; Cocoa Flavanols; Cocoa flavanols plus berries anthocyanins

SUMMARY:
The study examines the effect of cocoa flavanols, red-berries anthocyanins or a combination of both on markers of cardiovascular health and cognition.

DETAILED DESCRIPTION:
The study examines the effect of cocoa flavanols, red-berries anthocyanins or a combination of both on markers of cardiovascular health and cognition.

Healthy volunteers are recruited to participate in a parallel study (n 30 per group) for 10 to 12 weeks. Markers of cardiovascular health (FMD, markers of inflammation and fatty acid metabolism) and cognition (neuropsychological tests and plasma neurotrophins) are being measured before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-85
* BMI 20-32 Kg/m2

Exclusion Criteria:

* Mini-mental state examination (MMSE) < 28
* Systolic blood pressure (SBP) >139 mmHg
* Diastolic blood pressure (DBP) > 89 mmHg
* Total cholesterol > 6.5 mmol/L

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline of flow-mediated vasodilatation (FMD) of the brachial artery | Over 6 minutes on day 0 and after10 weeks
  The FMD of the brachial artery will be measured using an ultrasound collected at baseline and continuously for 60 seconds post-arm occlusion for 5 minutes. FMD will be expressed as percentage of variation between pre-and postischemic diameters

SECONDARY OUTCOMES:
Change from baseline STROOP score after 10 weeks intervention | at inclusion and 10 weeks after intervention
  STROOP tests attention and executive function. This test aims to evaluate the inhibition of an automated process such as reading by asking participants to name the color of color names written in a different color ink.
  For each participant SROOP results at inclusion will be compared with results after 10 weeks intervention
Change from baseline Tower of London score after 10 weeks intervention | at inclusion and 10 weeks after intervention
  Tower of London test consist of a three color game board that allows executive functioning evaluation by total time, time to first move and optimal moves change from participants inclusion to week 11.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Food Science, Technology and Nutrition (ICTAN), Spanish National Research Council (CISC), Madrid, Spain

IPD SHARING:
Plan to Share IPD: No